CLINICAL TRIAL: NCT06627153
Title: Epidemiological Assessment of Technical Diving Accidents in Mainland France and Factors Predictive of Severity
Brief Title: Epidemiological Assessment of Technical Diving Accidents in Mainland France and Factors Predictive of Severity (TEKCare)
Acronym: TEKCare
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0150 - TEKCare
Record Dates: First submitted 2024-09-23; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Decompression Sickness; Pulmonary Edema - Acute; Oxygen Toxicity; Carbon Dioxide Poisoning; Nitrogen Narcosis
MeSH Terms: conditions — Decompression Sickness; Inert Gas Narcosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims at an epidemiological description of the clinical presentation of medical problems in technical diving. It assess anthropometric data, diving experience and dive planification, clinical presentation, treatment received and pronostic to understand specificity of this community.

DETAILED DESCRIPTION:
In recent years, the increased availability of breathing gas mixtures, together with progressive technical development of specialized diving equipment, has contributed to expansion of the diver's community. Deep and long dives expose to decompression sickness (DCS) risk and hyperbaric oxygen therapy (HBO) is the definitive treatment. Incidence, clinical expression or prognosis of pathological events after technical diving might differ from recreational ones. A better knowledge of these specificity will facilitate risk assessment, analysis and medical care for hyperbaric physician community.

ELIGIBILITY:
Inclusion Criteria:

* Civilian technical diver
* Diving accident history (decompression sickness, biochemical accident or immersion pulmonary edema) following a technical dive in a trimix and/or rebreather dive
* Treated in a hyperbaric center on the coast of mainland France

Exclusion Criteria:

* Participation denied by the diver
* Diving incident diagnosis not retained by the hyperbaric physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Technical divers are defined by specialized equipment (e.g. rebreather) and/or helium based mixed-gases used to conduct deeper and longer dives. All divers who consulted hyperbaric installations after one of these dives with a retained diagnosis of a diving accident are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic description of injured technical divers treated in French hyperbaric center | 15 years
  Comparison of technical diver populations according to length of hospitalization (< 48 hours vs > 48 hours) corresponding to treatment with simple hyperbaric oxygen therapy or requiring several consolidation sessions in view of the severity and/or intensity of symptoms.

SECONDARY OUTCOMES:
Predictive factor of severity | 15 years
  Evaluation regarding the number of OHB treatment (reflecting the gravity if more than 2) and diving profil (breathing apparatus, maximal depth, dive total time, composition of mixed gas), demographic profile of divers (age, sex, medical conditions) and symptoms presentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement